CLINICAL TRIAL: NCT04142632
Title: Long Term Follow-up for Hypospadias. Hypospadias KOK
Brief Title: Long Term Follow-up for Hypospadias
Acronym: KOK
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0334; 2019-A02136-51 (Other: ID-RCB)
Record Dates: First submitted 2019-09-27; First posted 2019-10-29 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endocrinian sample: testosterone, FSH, LH, AMH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- long term evaluation of hypospadias surgery
  Interventions: Procedure: clinical and paraclinical examination

INTERVENTIONS:
Procedure: clinical and paraclinical examination — Physical examination of the penis, ultrasonography of the bladder end the testis, Biological sample for endocrine assessment

SUMMARY:
Hypospadias is a frequent malformation. The definition of hypospadias is a ventral tissues hypoplasia, with an abnormal position of the urethral meatus, a chordee of the penis and an open foreskin. It can be associate with other genital malformation; in that case it can be classified in the wider field of the disorder of sex development (DSD). There is a lot of surgical technics for those malformations.

In the pediatric surgical department, in Lyon, three technics are the most used because of their reliability and their good outcomes in short and mid term.

This is essential for investigator to have a long term evaluation, with a physical exam and paraclinical exams, after the puberty, to assess the outcomes after the changes especially at the puberty.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* with previous hypospadias surgery,
* Birthday before December the 31th 2009.
* The surgery was performed by one operator, with the following surgical technics: Koff, Onlay and Koyanagi.
* The patients are informed by an official surgery department letter, to assure they agree to participate.
* if the patient is still an infant, the parental agreement will be necessary.

Exclusion Criteria:

* Patient deceased
* Non- agreement from the patient or his parents
* Language difficulties

Min Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients with previous hypospadias surgery, the intervention has to be realized before December the 31th 2005.The surgery was performed by one operator (Pr MOURIQUAND), with the following surgical technics: Koff, Onlay and Koyanagi.
  The patients are informed by an official surgery department letter, to assure they agree to participate. If the patient is still an infant, the parental agreement will be necessary.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | Day 0
  Time with no complication after the last surgery for hypospadias

SECONDARY OUTCOMES:
Penis size | Day 0
Urinary symptoms | Day 0
  The investigator will do an interrogation of the patient about urinary symptoms, the response will be yes or no.
quality of the urinary flow: straight or not straight | Day 0
occurrence of urinary infection | Day 0
sexual activity | Day 0
  The investigator will do an interrogation of the patient about sexual activity, the response will be yes or no.
occurrence of ejaculation | Day 0
occurrence of erection | Day 0
Pre-voiding bladder volume | Day 0
post-voiding bladder volume | Day 0
Flow measurement | Day 0
  The investigator will use an urinary flowmeter; the investigator will collect data with a curve for each patient, with time in x-axis and ml/s in y-axis.
Testicular ultrasonography | day 0
  The investigator will ask a testicular ultrasonography which will be performed by a radiologist, the following data will be collected: testicular volume, aspect of the testicular parenchyma.
puberty clinical signs | Day 0
  The investigator will use the tanner's criteria during the physical examination.
  Stages of genital [G] and pubic hair [Ph] development in the male. G-1, Ph-1: pre-pubertal; G-2: the testis and scrotum enlarge, and the skin of the scrotum shows some reddening and change in the texture. Sparse growth of pigmented hair usually slightly curly, mainly at the base of the penis (Ph-2); G-3: Testis and scrotum enlarge further, the penis grows mainly in length but also in breadth. The hair is darker, coarser and curlier and spreads over the junction of the pubes (Ph-3); G-4: Scrotum, testis, and penis grow further with development of the glans, and further darkening of the scrotal skin. The hair spreads covering the pubes; G-5: adult stage with spreading of the hair to the medial surface of the thighs (Ph-5).
endocrine disorder | Day 0
patient satisfaction | day 0
  The investigator will do an interrogation of the patient about his personal satisfaction, the response will be yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Valeska BIDAULT, MD, Principal Investigator — Hospices Civils de Lyon Service de chirurgie uro-viscérale, thoracique et de transplantation de l'enfant Hôpital Femme Mère Enfant
Locations (1):
- Service de chirurgie uro-viscérale, thoracique et de transplantation de l'enfant Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No